CLINICAL TRIAL: NCT04516265
Title: The Comparison of Effectiveness of Structured Trunk Training Protocols in Patients With Cerebral Palsy
Brief Title: Effects of Trunk Training in Patients With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Derya Azim Rezaei, lecturer, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Okan U
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Cerebral Palsy
Keywords: trunk training; theratogs; exercise game; video-based training
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Patients with cerebral palsy will be divided into 3 groups in a randomized controlled manner. Each group will continue and follow routine physiotherapy and rehabilitation treatments for 8 weeks. Then, structured trunk training will begin. NGT-based trunk training (45 minutes) to the first group, video-based trunk training (45 minutes) to the second group, and Video-based trunk training (45 minutes) will apply with Theratogs to the third group. Treatments will be applied two days a week for 8 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NGT Group (Active Comparator): A personally designed treatment program will be applied in line with the principles of neurodevelopmental treatment.
  Interventions: Procedure: neurodevelopmental treatment
- Video-based training group (Active Comparator): Trunk training will be done with games developed for the use of children with cerebral palsy.
  Interventions: Procedure: video-based trunk training
- Video-based training group with theratogs (Active Comparator): Video-based trunk training (45 minutes) will apply with Theratogs to the group
  Interventions: Procedure: Video-based trunk training will apply with Theratogs

INTERVENTIONS:
Procedure: neurodevelopmental treatment — A personally designed treatment program will be applied in line with the principles of neurodevelopmental treatment.
  Arms: NGT Group
Procedure: video-based trunk training — Games developed for the use of children with cerebral palsy will be used for trunk training.
  Arms: Video-based training group
Procedure: Video-based trunk training will apply with Theratogs — Video-based trunk training will apply with Theratogs
  Arms: Video-based training group with theratogs

SUMMARY:
The aim of our study is to compare the effects of NGT-based trunk training, video-based trunk training and video-based trunk training applied with Theratogs in children with hemiparetic type Cerebral Palsy.

DETAILED DESCRIPTION:
The aim of our study is to compare the effects of NGT-based trunk training, video-based trunk training and video-based trunk training applied with Theratogs in children with hemiparetic type Cerebral Palsy. It is planned to include 45 patients with hemiparetic cerebral palsy between the ages of 5-15 and with Gross Motor Function Classification System (GMFCS) level I-III. Patients with cerebral palsy will be divided into 3 groups in a randomized controlled manner. Each group will continue and follow routine physiotherapy and rehabilitation treatments for 8 weeks. Then, structured trunk training will begin. NGT-based trunk training (45 minutes) to the first group, video-based trunk training (45 minutes) to the second group, and Video-based trunk training (45 minutes) will apply with Theratogs to the third group. Treatments will be applied two days a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with I-III levels according to Communication Function Classification System
* Patients with I-III levels according to GMFCS
* Patients with Hemiparetic Cerebral Palsy
* Continuing regular physiotherapy and rehabilitation program for six months.

Exclusion Criteria:

* Presence of visual or auditory impairment
* Presence of epilepsy
* Patients who have undergone orthopedic surgery in the last 6 months
* Patients who received Botulinum Toxin-A injection in the last 6 months

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-07-21 (Estimated); Study Completion 2021-09-21 (Estimated)

PRIMARY OUTCOMES:
Trunk Control Measurement Scale | 8 weeks
  It will be used to evaluate trunk control in patients with CP.
Trunk Muscle Tone | 8 weeks
  Trunk Muscle Tone will be evaluated with the Myoton®PRO device.
Segmental Assesment of Trunk Control Scale | 8 weeks
  It is an evaluation method that allows the body control to be evaluated from 3 different aspects as static, active and reactive control, according to trunk control levels.
Balance Assessment System | 8 weeks
  The Fizyosoft Balance Assessment system, which works in harmony with the Nintendo Wii Balance Board, will be used in the assessment of the sitting balance.

SECONDARY OUTCOMES:
Pediatric Berg Balance Scale | 8 weeks
  It will be used to assess functional balance.
10-meters walking test | 8 weeks
  It will be used to evaluate walking.
Gillette Functional Gait Assessment Questionaire | 8 weeks
  It will be used to evaluate functional walking.

CONTACTS AND LOCATIONS:
Overall Officials: Derya Azim Rezaei, MSc, Principal Investigator — Okan University,Faculty of Health Sciences,Department of Physiotherapy and Rehabilitation; Burcu Ersöz Hüseyinsinoğlu, Associate professor, Study Director — Istanbul University-Cerrahpaşa,Faculty of Health Sciences,Department of Physiotherapy and Rehabilitation
Locations (1):
- Okan University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No